CLINICAL TRIAL: NCT00394290
Title: Follow-up of the Therapeutic Coverage by Continuous Positive Pressure of the Obstructive Sleep Apnea Syndrome for Down Syndrome Patients
Brief Title: Down Syndrome and Continuous Positive Pressure Therapy
Acronym: Morphee
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Jerome Lejeune (Other)
Collaborators: Fondation Jérôme Lejeune (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IJL-PPC-EP02; Morphee
Record Dates: First submitted 2006-10-31; First posted 2006-11-01 (Estimated); Last update posted 2019-03-26 (Actual); Status verified 2012-10

CONDITIONS: Down Syndrome; Obstructive Sleep Apnea Syndrome
Keywords: Down Syndrome; Obstructive Sleep Apnea Syndrome; Continuous Positive Pressure; Hypersomnia
MeSH Terms: conditions — Down Syndrome; Sleep Apnea, Obstructive; Disorders of Excessive Somnolence | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- PPC (Experimental): Night time device for positive pulmonary pressure
  Interventions: Device: Continuous Positive Pressure

INTERVENTIONS:
Device: Continuous Positive Pressure — Nighttime continuous positive pressure device, to be used every day

SUMMARY:
The purpose of this study is to evaluate the efficacy and tolerability of Continuous Positive Pressure for SAOS in Down Syndrome patients.

ELIGIBILITY:
Inclusion Criteria:

* Down Syndrome patients with an Obstructive Sleep Apnea Syndrome
* more than 18 years old

Exclusion Criteria:

* predictable non-compliance of device
* non-compensated cardiopathy
* non-stable thyroxin treatment
* non-stable diabetes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2006-11-16 (Actual); Primary Completion 2012-10-31 (Actual); Study Completion 2012-12-31 (Actual)

PRIMARY OUTCOMES:
Scores on psychometrical and dementia scales after a 3-month treatment period (and if possible, after 12 months) | 0 and 3 months

SECONDARY OUTCOMES:
Tolerability | 0, 3 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Martine Conte, M.D., Principal Investigator — Institut Jerome Lejeune; Franck STURTZ, M.D., Study Director — Institut Jerome Lejeune
Locations (1):
- Institut Jerome Lejeune, Paris, France

REFERENCES:
- [Background] Resta O, Barbaro MP, Giliberti T, Caratozzolo G, Cagnazzo MG, Scarpelli F, Nocerino MC. Sleep related breathing disorders in adults with Down syndrome. Downs Syndr Res Pract. 2003 Aug;8(3):115-9. doi: 10.3104/reports.138. PMID 14502839